CLINICAL TRIAL: NCT05055778
Title: Establishing the Effectiveness of Publicly Available Smoking Cessation Resources: Does Rurality Matter?
Brief Title: Establishing the Effectiveness of Publicly Available Smoking Cessation Resource
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Kara Wiseman, MPH, PhD, Assistant Professor, Department of Public Health Sciences, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3928
Record Dates: First submitted 2021-08-16; First posted 2021-09-24 (Actual); Results first posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SmokfreeTXT (Experimental): Research version of the publicly available SmokefreeTXT program
  Interventions: Behavioral: SmokefreeTXT

INTERVENTIONS:
Behavioral: SmokefreeTXT — The program is identical to the publicly available program available through the National Cancer Institute Smokefree.gov Initiative but has been set up to be delivered through a research account. The program will send 3-5 messages a day over 7 weeks, with one week to prepare for a quit attempt and 6 weeks of cessation support messages. Participants can get real time support for cravings, mood, and slips by texting "keywords" to the program. They keywords are CRAVE, MOOD, and SLIP. Participants can also re-set their quit date by texting NEW. The program asks questions each week to ask about smoking status and about mood and cravings.

SUMMARY:
The purpose of this study is to evaluate the effectiveness of SmokefreeTXT, a smoking cessation text messaging program currently available to anyone in the United States through www.smokefree.gov, and to compare cessation outcomes for smokers living in different regions of Virginia while participants use the program. Participants will be asked to complete assessments at Baseline, 7 weeks, 3 months, and 6 months and will be asked to use a research version of SmokefreeTXT.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and over
* Current cigarette smoker (has smoked at least 100 cigarettes in their lifetime and currently smokes)
* Ability to read and speak English
* Resident of Virginia
* Owns a cell phone

Exclusion Criteria:

* Not a current smoker (e.g., started a quit attempt between providing interest information and starting the study)
* Identity not able to be verified from information provided on interest form
* Does not own a cell phone
* Pregnant smoker or may become pregnant in the next 6 months
* Lives in an area that has met recruitment criteria (after recruitment has begun)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2021-11-03 (Actual); Primary Completion 2024-02-06 (Actual); Study Completion 2024-02-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
If requested, a de-identified dataset will be available to other researchers after the study is completed.
Supporting Information: Study Protocol
Time Frame: After study completion

REFERENCES:
- [Derived] Kinchen JW, Little MA, Ritterband LM, Wiseman KP. Pilot study examining the effect of rurality on engagement and abstinence for adult users of a text-message cessation intervention. BMC Public Health. 2025 Nov 19;25(1):4061. doi: 10.1186/s12889-025-25284-6. PMID 41257752

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SmokfreeTXT
Started | 49
Completed | 49
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | SmokfreeTXT
Number analyzed (Participants) | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.3 (11.9)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 6
  Female | 41
  Censored | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 36
  Non-Hispanic Black | 7
  Other | 6
Region of Enrollment [Number; unit: participants]
  United States | 49
Daily smoking status [Count of Participants; unit: Participants]
  Every day | 44
  Some days | 5
County-level rurality [Count of Participants; unit: Participants]
  Rural (RUCA 4-10) | 23
  Non-Rural (RUCA 1-3) | 26

OUTCOME MEASURES:

1. Primary Outcome: Self-reported Smoking Cessation
Description: 7-day point prevalence of abstinence (Question wording: Have you smoked a cigarette (even a puff) in the past 7 days? Response options: Yes; No)
Time Frame: 7 weeks after study start
Population: Non-responders coded as continuing to smoke
Measure: Count of Participants; unit: Participants
Arm/Group | SmokfreeTXT
Number analyzed (Participants) | 49
Participants | 16

2. Primary Outcome: Self-reported Smoking Cessation
Description: as for outcome 1
Time Frame: 3 months
Population: Non-responders coded as continuing to smoke
Measure: Count of Participants; unit: Participants
Arm/Group | SmokfreeTXT
Number analyzed (Participants) | 49
Participants | 14

3. Secondary Outcome: Self-reported Continuous Abstinence
Description: Continuous abstinence, 6 weeks after initiating the quit attempt (Question wording: In the last 6 weeks, have you smoked at all? Response options: Yes; No; Not sure)
Time Frame: 7 weeks after study start
Population: Participants who did not respond are coded as continuing to smoke
Measure: Count of Participants; unit: Participants
Arm/Group | SmokfreeTXT
Number analyzed (Participants) | 49
Participants
  Yes | 42
  No | 6
  Not Sure | 1

4. Secondary Outcome: Self-reported Continuous Abstinence
Description: Continuous abstinence 3 months after initiating the quit attempt (Question wording: In the last 3 months, have you smoked at all? Response options: Yes; No; Not sure)
Time Frame: 3 months
Population: Non-responders coded as continuing to smoke
Measure: Count of Participants; unit: Participants
Arm/Group | SmokfreeTXT
Number analyzed (Participants) | 49
Participants
  Yes | 43
  No | 6
  Not Sure | 0

5. Secondary Outcome: Self-reported Smoking Cessation
Description: as for outcome 1
Time Frame: 6 months
Population: Non-responders coded as continuing to smoke
Measure: Count of Participants; unit: Participants
Arm/Group | SmokfreeTXT
Number analyzed (Participants) | 49
Participants | 18

6. Secondary Outcome: Self-reported Continuous Abstinence
Description: Continuous abstinence 6 months after initiating the quit attempt (Question wording: In the last 6 months, have you smoked at all? Response options: Yes; No; Not sure)
Time Frame: 6 months
Population: Any participants who did not respond to the 6-month survey was coded as continuing to smoke.
Measure: Count of Participants; unit: Participants
Arm/Group | SmokfreeTXT
Number analyzed (Participants) | 49
Participants
  Yes | 43
  No | 6
  Not Sure | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over 6 months from time of enrollment for each participant
Arm/Group | SmokfreeTXT
All-Cause Mortality (participants affected / at risk) | 0/49
Serious Adverse Events (participants affected / at risk) | 0/49
Other Adverse Events (participants affected / at risk) | 0/49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-25): https://cdn.clinicaltrials.gov/large-docs/78/NCT05055778/Prot_SAP_000.pdf